CLINICAL TRIAL: NCT06012994
Title: Retrospective Study of the Protective Effect of Gastrodin on Myocardium in Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: mzk202303
Record Dates: First submitted 2023-08-20; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GAS
- Control

SUMMARY:
Retrospective collection of Wuhan Union hospital from December 1,2018 to June 30,2021 to meet the entry and discharge standards. The patient 's medical record data were divided into study group and control group according to the use of gastrodin during operation. The perioperative data and prognostic outcomes in the patient 's medical records were collected and analyzed. The degree of myocardial injury and postoperative clinical outcomes were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged≥18 years, regardless of gender;
* Patients undergoing elective cardiac surgery under general anesthesia;
* ASA grade 1 ~ 3.

Exclusion Criteria:

* Suffering from more serious genetic diseases (such as immunodeficiency, thalassemia, etc.);
* Moderate to severe malnutrition, moderate to severe anemia;
* Persistent infection;
* Severe preoperative underlying diseases (such as severe liver and kidney dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included patients who were preoperatively diagnosed as requiring elective thoracic cardiac surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The degree of myocardial injury | The myocardial tissue was collected during the operation. About 2 hours on average
  The myocardial tissue trimmed by the surgeon according to the surgical requirements was collected during the operation for electron microscopy observation and detection of related molecular content.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China